CLINICAL TRIAL: NCT00640445
Title: Military to Civilian: RCT of an Intervention to Promote Postdeployment Reintegration
Brief Title: Military to Civilian: Trial of an Intervention to Promote Postdeployment Reintegration
Acronym: M2C
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Nina A. Sayer, Associate Director, CCDOR; Research Director, PTBRI QUERI, Minneapolis Veterans Affairs Medical Center
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: PT074432
Record Dates: First submitted 2008-03-18; First posted 2008-03-21 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Clinical Trial; Combat Disorders; PTSD; Internet-Based Intervention; Mental Health Services; Post-deployment Reintegration
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Combat Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Expressive Writing (Experimental): Participants assigned to the Expressive Writing (EW) condition will write about their deepest thoughts and feelings associated with their experience transitioning from being a soldier to being a civilian for 20 minutes a day for 4 days within a week.
  Interventions: Behavioral: Expressive Writing
- Control Writing (Active Comparator): Those assigned to control writing condition will write factually about the information needs of veterans transitioning from active duty to civilian status for 20 minutes on 4 days within one week.
  Interventions: Behavioral: Control Writing
- No Writing Control (No Intervention): Treatment As Usual

INTERVENTIONS:
Behavioral: Expressive Writing — In EW, people are asked to write about their deepest thoughts and feelings surrounding a significant life event for 20 minutes a day for 4 days
  Arms: Expressive Writing
Behavioral: Control Writing — Those assigned to control writing conditions are asked to describe factual information for 20 minutes a day for 4 days.
  Arms: Control Writing

SUMMARY:
Veterans returning from combat deployments face the interrelated challenges of processing their combat experiences and transitioning back to civilian life. Unfortunately, many veterans wait years or decades before seeking help for post-deployment problems, if they seek it at all. This study seeks to determine whether Internet-Based Expressive Writing (IB-EW), a brief, low-cost, easily disseminated, and resource-efficient intervention, can reduce psychological symptoms and improve functioning among Operation Iraqi Freedom (OIF) and Operation Enduring Freedom (OEF) veterans as they navigate this transition, while also attempting to reduce barriers to help-seeking. Expressive Writing, a highly private, readily accessible, and non-stigmatizing intervention, has a strong evidence-base in civilian populations, but its efficacy in combat veterans has not been tested. This study therefore seeks to test the efficacy of Expressive Writing in a veteran population while further enhancing its accessibility by delivering it over the internet (Internet-Based Expressive Writing; IB-EW). This study will comprise a randomized controlled trial with three conditions: (a) Internet-Based Expressive Writing, (b) Internet-Based Control Writing, and (c) No Writing/Treatment As Usual, with a total of 1152 OIF/OEF veterans randomized across these groups. Expressive Writing participants will write with feeling about their transition from being a soldier to being a civilian; Control Writing participants will write factually about the information needs of new veterans; and Treatment as Usual participants will complete the assessments but not engage in any writing assignments. Participants will complete standardized self-report measures of psychological symptoms, psychosocial functioning, and life satisfaction at baseline (Session 1) and at three months (Session 6) and six months (Session 7) post-intervention. Participants in writing conditions will write for 20 minutes on four consecutive days (Sessions 2-5) following completion of baseline measures (participants in the TAU condition will not complete Sessions 2-5). The study will also attempt to identify individual difference characteristics related to the efficacy of the treatment, to see who may be most likely to benefit from the treatment. Analyses will primarily entail multivariate analyses of variance. Power is adequate to detect even a small effect.

ELIGIBILITY:
Inclusion Criteria:

* Veteran from current wars in Iraq and Afghanistan
* At least a little difficulty transitioning from soldier to civilian
* Access to computer with internet
* Provide valid contact information
* Available to participate for up to 40 minutes per session
* Interested in participation
* Understand procedures and consent
* Note: participants are recruited by random selection from the target population

Exclusion Criteria:

* Severe depression

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1292 (Actual)
Dates: Start 2011-06; Primary Completion 2013-04 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
PTSD symptoms | Baseline, 3-month, 6-month
Hostility | Baseline, 3-month, 6-month
Psychological distress | Baseline, 3-month, 6-month
Physical symptoms | Baseline, 3-month, 6-month
Reintegration difficulty | Baseline, 3-month, 6-month
Social support | Baseline, 3-month, 6-month
Life satisfaction | Baseline, 3-month, 6-month

SECONDARY OUTCOMES:
Emotion and causal word use in participants' essays | Intervention Sessions (up to 4 sessions post-baseline for participants assigned to a writing condition)
Employment status | Baseline, 3-month, 6-month

CONTACTS AND LOCATIONS:
Overall Officials: Nina A Sayer, PhD, Principal Investigator — Minneapolis Veterans Affairs Medical Center
Locations (1):
- VA Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Sayer NA, Orazem RJ, Noorbaloochi S, Gravely A, Frazier P, Carlson KF, Schnurr PP, Oleson H. Iraq and Afghanistan War Veterans with Reintegration Problems: Differences by Veterans Affairs Healthcare User Status. Adm Policy Ment Health. 2015 Jul;42(4):493-503. doi: 10.1007/s10488-014-0564-2. PMID 24913102